CLINICAL TRIAL: NCT04422808
Title: Assessing Current Analgesia and Sedation Weaning Practices in Adult Critically Ill Patients
Brief Title: AduLt iatrogEnic withdRawal sTudy in the ICU (ALERT-ICU)
Status: Completed | Type: Observational
Sponsor: Wilkes University (Other)
Responsible Party: Principal Investigator, Scott Bolesta, Pharm.D., BCPS, FCCM, FCCP, Associate Professor, Wilkes University
Other Study IDs: 116
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Withdrawal Syndrome; Iatrogenic Disease
Keywords: Opioid withdrawal; Benzodiazepine withdrawal; Narcotic withdrawal; Critically ill
MeSH Terms: conditions — Substance Withdrawal Syndrome; Iatrogenic Disease; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Withdrawal from opioids and sedatives administered for medical purposes (i.e. iatrogenic withdrawal) often goes unrecognized in the critically ill, but its prevalence is high. Reports describing what is being implemented at the bedside to prevent iatrogenic withdrawal are lacking, and how patients are monitored and assessed for withdrawal has not been adequately studied. Therefore, the investigators overall objective is to determine the current analgesia and sedation weaning practices in adult ICUs. In order to accomplish this objective the investigators plan to conduct a prospective, observational, point prevalence trial. Data from this project will help support future investigation of iatrogenic withdrawal.

DETAILED DESCRIPTION:
The design for this study will be an international, prospective, observational, point prevalence trial. The investigators plan to recruit multiple sites to participate in the study through the use of professional organization list serves as well as direct outreach to colleagues and associates of members of the investigator team. Data collection will be performed by site investigators on one single day for all patients currently in the ICU who meet inclusion criteria on the data collection day. Site investigators will have an approximately three-month time frame in which to choose a data collection date. All data collection will be performed using REDcap, a secure web-based data collection tool that meets the HIPAA (Health Insurance Portability and Accountability Act of 1996) requirements for protection of patient health information. Utilization of this system will allow real-time input of data from the patient's bedside by site investigators. Data collected will include various site and patient demographic data. The investigators will also collect opioid and sedative doses, durations of therapy, weaning of doses, and withdrawal assessment results.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years and older admitted to an adult intensive care unit on the day of data collection who have received parenteral analgesics or sedatives in the previous 24 hours.

Exclusion Criteria:

* Patients who have not received parenteral analgesics or sedatives in the previous 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We anticipate the involvement of at least 50 intensive care unit centers within the United States, and less than 10 sites outside the United States (primarily in Canada, Australia, Europe, and the Middle East). Estimating an average of 10 patients who meet study criteria at each site.
Sampling Method: Non-Probability Sample
Enrollment: 2437 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Number patients weaned from parenteral analgesics | Three months
  The primary outcome will be the number of patients who are weaned from continuous parenteral analgesics and sedatives using a standardized approach. Continuous analgesic and sedative administration will be defined as those given as a continuous intravenous infusion, scheduled intermittent intravenous or subcutaneous injections, or as needed with at least half of the possible doses in a 24 hour period being administered.

SECONDARY OUTCOMES:
Patient proportion | Three months
  Proportion of ICU patients who are receiving continuous analgesics and sedatives
Utilized analgesic and sedative weaning practice | three months
  Types of analgesic and sedative weaning practices being utilized in adult ICU patients.
Number of patients assessed | three months
  Number of patients being assessed for iatrogenic withdrawal after receiving continuous analgesics and sedatives.
Assessment tools | three months
  Assessment tools being utilized for iatrogenic withdrawal.
Standardized approach patients | three months
  Number of patients in which a standardized approach to iatrogenic withdrawal assessment is being utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles L Fraser, PharmD, MCCM, Study Director — Tufts University School of Medicine; Scott Bolesta, PharmD, BCPS, Principal Investigator — Wilkes University; Marc M Perreault, MSc, PharmD, Study Director — Université de Montréal; Lisa Burry, PharmD, Study Director — MOUNT SINAI HOSPITAL; Brian L Erstad, PharmD, MCCM, Study Director — The University of Arizona College of Pharmacy; Céline Gélinas, N., Ph.D., Study Director — Ingram School of Nursing; Richard R Riker, MD, FCCM, Study Director — Tufts University School of Medicine; Katrianna D Saltarelli, Student, Study Chair — Wilkes University; Jennifer Mitchell, Student, Study Chair — Wilkes University; Kathryn E Smith, PharmD, BCPS, BCCCP, Study Director — MaineHealth; Federico Carini, MD, Study Director — Hospital Italiano de Buenos Aires; Rebekah Eadie, MPharm, MSc, IP, MPSNI, Study Director — Ulster Hospital- South Eastern Health and Social Care Board; Jamie Harpel, Student, Study Chair — Wilkes University; Ryan Stewart, Student, Study Chair — Wilkes University
Locations (1):
- Wilkes University, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to share individual participant data specific to each institution through data access groups in RedCap
Supporting Information: Study Protocol, SAP
Time Frame: Twelve months after data collection completed.
Access Criteria: Individual site data will be accessible to each specific participating study site. Only site investigators will have access to their study site data.

REFERENCES:
- [Result] Borkowska M, Labeau S, Schepens T, Vandijck D, Van de Vyver K, Christiaens D, Lizy C, Blackwood B, Blot SI. Nurses' Sedation Practices During Weaning of Adults From Mechanical Ventilation in an Intensive Care Unit. Am J Crit Care. 2018 Jan;27(1):32-42. doi: 10.4037/ajcc2018959. PMID 29292273
- [Result] Brown C, Albrecht R, Pettit H, McFadden T, Schermer C. Opioid and benzodiazepine withdrawal syndrome in adult burn patients. Am Surg. 2000 Apr;66(4):367-70; discussion 370-1. PMID 10776874
- [Result] Cammarano WB, Pittet JF, Weitz S, Schlobohm RM, Marks JD. Acute withdrawal syndrome related to the administration of analgesic and sedative medications in adult intensive care unit patients. Crit Care Med. 1998 Apr;26(4):676-84. doi: 10.1097/00003246-199804000-00015. PMID 9559604
- [Result] Chiu AW, Contreras S, Mehta S, Korman J, Perreault MM, Williamson DR, Burry LD. Iatrogenic Opioid Withdrawal in Critically Ill Patients: A Review of Assessment Tools and Management. Ann Pharmacother. 2017 Dec;51(12):1099-1111. doi: 10.1177/1060028017724538. Epub 2017 Aug 9. PMID 28793780
- [Result] Curley MA, Wypij D, Watson RS, Grant MJ, Asaro LA, Cheifetz IM, Dodson BL, Franck LS, Gedeit RG, Angus DC, Matthay MA; RESTORE Study Investigators and the Pediatric Acute Lung Injury and Sepsis Investigators Network. Protocolized sedation vs usual care in pediatric patients mechanically ventilated for acute respiratory failure: a randomized clinical trial. JAMA. 2015 Jan 27;313(4):379-89. doi: 10.1001/jama.2014.18399. PMID 25602358
- [Result] Duceppe MA, Perreault MM, Frenette AJ, Burry LD, Rico P, Lavoie A, Gelinas C, Mehta S, Dagenais M, Williamson DR. Frequency, risk factors and symptomatology of iatrogenic withdrawal from opioids and benzodiazepines in critically Ill neonates, children and adults: A systematic review of clinical studies. J Clin Pharm Ther. 2019 Apr;44(2):148-156. doi: 10.1111/jcpt.12787. Epub 2018 Dec 19. PMID 30569508
- [Result] Fonsmark L, Rasmussen YH, Carl P. Occurrence of withdrawal in critically ill sedated children. Crit Care Med. 1999 Jan;27(1):196-9. doi: 10.1097/00003246-199901000-00052. PMID 9934916
- [Result] Wang PP, Huang E, Feng X, Bray CA, Perreault MM, Rico P, Bellemare P, Murgoi P, Gelinas C, Lecavalier A, Jayaraman D, Frenette AJ, Williamson D. Opioid-associated iatrogenic withdrawal in critically ill adult patients: a multicenter prospective observational study. Ann Intensive Care. 2017 Sep 2;7(1):88. doi: 10.1186/s13613-017-0310-5. PMID 28866754
- [Derived] Bolesta S, Burry L, Perreault MM, Gelinas C, Smith KE, Eadie R, Carini FC, Saltarelli K, Mitchell J, Harpel J, Stewart R, Riker RR, Fraser GL, Erstad BL; AduLt iatrogEnic withdRawal sTudy in the ICU (ALERT-ICU) Study Investigators. International Analgesia and Sedation Weaning and Withdrawal Practices in Critically Ill Adults: The Adult Iatrogenic Withdrawal Study in the ICU. Crit Care Med. 2023 Nov 1;51(11):1502-1514. doi: 10.1097/CCM.0000000000005951. Epub 2023 Jun 7. PMID 37283558